CLINICAL TRIAL: NCT05126303
Title: A Phase 2, Randomized, Placebo-Controlled, Double-Blind, Adaptive, Parallel Group Clinical Study to Evaluate the Efficacy and Safety of RMC-035 in Subjects at High Risk for Acute Kidney Injury Following Open-Chest Cardiac Surgery
Brief Title: Efficacy and Safety of RMC-035 in Subjects at High Risk for Acute Kidney Injury Following Open-Chest Cardiac Surgery
Acronym: AKITA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment discontinued following DMC recommendation based on futility with regards to primary endpoint
Sponsor: Guard Therapeutics AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 21-ROS-05
Record Dates: First submitted 2021-11-08; First posted 2021-11-19 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, adaptive, parallel group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- RMC-035 (Experimental): RMC-035 is a concentrate (6.0 mg/mL) for solution for infusion for IV administration.
  Dosing will be based on renal function at Day -1: Subjects with eGFR ≥60 mL/min/1.73m2 will receive 1.3 mg/kg (per dose) for the first and second dose, followed by 0.65 mg/kg (per dose) for the third, fourth and fifth dose, while subjects with eGFR >30 and <60 mL/min/1.73m2 will receive 0.65 mg/kg (per dose) for all five doses Dosing occurs at time 0 and then after 6, 12, 24 and 48 hours.
  Interventions: Drug: RMC-035
- Placebo (Placebo Comparator): Identical to RMC-035 arm except that the placebo contains no active ingredient.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RMC-035 — Concentrate for Solution for Infusion
  Other Names: ROSgard
  Arms: RMC-035
Drug: Placebo — Concentrate for Solution for Infusion
  Arms: Placebo

SUMMARY:
This study evaluates RMC-035 compared to placebo for the prevention of acute kidney injury (AKI) in subjects who are at high risk for AKI following cardiac surgery. Half of the subjects will receive RMC-035 and the other half will receive placebo.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind, adaptive, parallel group clinical study that will evaluate RMC-035 compared to placebo in subjects at high risk for acute kidney injury (AKI) following cardiac surgery. Subjects are randomized in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Institutional Review Board/ International Ethics Committee approved Informed Consent obtained
2. Ability to understand and comply with the study requirements and able to provide written informed consent
3. Age ≥18 and <85 years
4. Estimated glomerular filtration rate (eGFR) is ≥30 mL/min/1.73 m2
5. Subject is scheduled for non-emergent coronary artery bypass grafting (CABG) surgery and/or valve surgery and/or ascending aorta aneurysm surgery with use of cardiopulmonary bypass (CPB), and AKI risk factors are present at screening
6. Female subject is not of child-bearing potential, or agreeing not to become pregnant
7. Female subject must not be breastfeeding
8. Female subject must not donate ova
9. Male subject and their female spouse/partner(s) who are of childbearing potential must be using a highly effective form of birth control
10. Male subjects must not donate sperm
11. Subject agrees not to participate in another interventional study

Exclusion Criteria:

1. Medical condition that makes the subject unsuitable for study participation
2. Scheduled for emergent surgeries (eg, aortic dissection)
3. Scheduled for CABG and/or valve surgery and/or ascending aorta aneurysm surgery combined with additional non-emergent cardiac surgeries (eg, congenital heart defects)
4. Scheduled to undergo transcatheter aortic valve implantation (TAVI) or transcatheter aortic valve replacement (TAVR), or off-pump surgeries or left ventricular assist device (LVAD) implantation
5. Experiences a cardiogenic shock or hemodynamic instability which require inotropes or vasopressors or other mechanical devices within 24 hours prior to surgery
6. Requirement for defibrillator or permanent pacemaker, mechanical ventilation, intraaortic balloon pumping (IABP), LVAD, or other forms of mechanical circulatory support (MCS)
7. Diagnosed with AKI (as defined by KDIGO criteria) within 3 months prior to surgery
8. Required cardiopulmonary resuscitation within 14 days prior to cardiac surgery
9. Ongoing sepsis or an untreated diagnosed clinically significant infection (viral or bacterial)
10. Total bilirubin or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 2 times the upper limit of normal (ULN)
11. History of solid organ transplantation
12. History of renal replacement therapy (RRT)
13. Medical condition which requires active immunosuppressive treatment
14. Severe allergic asthma
15. Ongoing chemotherapy or radiation therapy for malignancy that may have an impact on kidney function
16. Received an investigational medicinal product within the last 90 days (or within 5 half-lives of the investigational drug, whichever is longer)
17. Subject has a known allergy to RMC-035 or one of its constituents, or has previously received RMC-035

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Agervald, MD, Study Director — Guard Therapeutics; Alexander Zarbock, MD, Principal Investigator — Muenster University Hospital
Locations (29):
- United States (8):
  - Indiana Ohio Heart, Fort Wayne, Indiana
  - Bryan Heart, Lincoln, Nebraska
  - Rochester Regional Health - Rochester General Hospital, Rochester, New York
  - Duke University Hospital, Durham, North Carolina
  - Baylor Scott and White Research Institute - Dallas, Dallas, Texas
  - University of Virginia (UVA) Health - University Hospital, Charlottesville, Virginia
  - University of Wisconsin, Madison, Wisconsin
  - Aurora Health Care - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Canada (6):
  - Hamilton Health Sciences, Hamilton
  - CHUM, Montreal
  - MUHC - Royal Victoria Hospital, Montreal
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec
  - St. John Regional Hospital, Saint John
  - Saint Michael's Hospital, Toronto
- Czechia (2):
  - University Hospital Hradec Kralove, Hradec Králové
  - University Hospital Motol - Charles University Prague, Prague
- Germany (8):
  - Herz- und Diabeteszentrum Nordrhein-Westfalen (NRW), Bad Oeynhausen
  - Universitätsklinikum Köln, Cologne
  - Herzzentrum Dresden GmbH, Dresden
  - Westdeutsches Herzzentrum Essen, Essen
  - Universitätsklinikum Giessen und Marburg - Standort Giessen, Giessen
  - Universitätsklinikum Halle (Saale), Halle
  - Deutsches Herzzentrum München, München
  - Münster University Hospital, Münster
- Spain (5):
  - Hospital Sant Pau, Barcelona
  - Reina Sofia University Hospital, Córdoba
  - Hospital de La Princesa, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Complejo Hospitalario Universitario de Santiago (CHUS), Santiago de Compostela

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zarbock A, Larsson TE, Noiseux N, Mazer CD, Bohm J, Laflamme M, Matschke K, Burkert J, de Varennes B, Myjavec A, Boning A, Koyner JL, Engelman D, Reusch M, Thielmann M; AKITA investigators. Efficacy and safety of therapeutic alpha-1-microglobulin RMC-035 in reducing kidney injury after cardiac surgery: a multicentre, randomised, double-blind, parallel group, phase 2a trial. EClinicalMedicine. 2024 Sep 16;76:102830. doi: 10.1016/j.eclinm.2024.102830. eCollection 2024 Oct. PMID 39318788
- [Derived] Mazer CD, Siadati-Fini N, Boehm J, Wirth F, Myjavec A, Brown CD, Koyner JL, Boening A, Engelman DT, Larsson TE, Renfurm R, de Varennes B, Noiseux N, Thielmann M, Lamy A, Laflamme M, von Groote T, Ronco C, Zarbock A. Study protocol of a phase 2, randomised, placebo-controlled, double-blind, adaptive, parallel group clinical study to evaluate the efficacy and safety of recombinant alpha-1-microglobulin in subjects at high risk for acute kidney injury following open-chest cardiac surgery (AKITA trial). BMJ Open. 2023 Apr 6;13(4):e068363. doi: 10.1136/bmjopen-2022-068363. PMID 37024249

RESULTS

PARTICIPANT FLOW:
Groups:
- RMC-035: RMC-035 is a concentrate (6.0 mg/mL) for solution for infusion for IV administration.
  Dosing was based on renal function on Day -1: Subjects with eGFR ≥60 mL/min/1.73m2 received 1.3 mg/kg (per dose) for the first and second dose, followed by 0.65 mg/kg (per dose) for the third, fourth and fifth dose, while subjects with eGFR >30 and <60 mL/min/1.73m2 received 0.65 mg/kg (per dose) for all five doses Dosing occurred at time 0 and then after 6, 12, 24 and 48 hours.
  RMC-035: Concentrate for Solution for Infusion
Period: Overall Study
Arm/Group | RMC-035 | Placebo
Started | 89 | 88
Completed | 89 | 88
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All dosed
Groups:
- RMC-035: RMC-035 is a concentrate (6.0 mg/mL) for solution for infusion for IV administration.
  Dosing was based on renal function at Day -1: Subjects with eGFR ≥60 mL/min/1.73m2 received 1.3 mg/kg (per dose) for the first and second dose, followed by 0.65 mg/kg (per dose) for the third, fourth and fifth dose, while subjects with eGFR >30 and <60 mL/min/1.73m2 received 0.65 mg/kg (per dose) for all five doses Dosing occurred at time 0 and then after 6, 12, 24 and 48 hours.
  RMC-035: Concentrate for Solution for Infusion
- Total: Total of all reporting groups
Arm/Group | RMC-035 | Placebo | Total
Number analyzed (Participants) | 89 | 88 | 177
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 17 | 36
  >=65 years | 70 | 71 | 141
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 70 | 69 | 139
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 82 | 81 | 163
  Unknown or Not Reported | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 86 | 85 | 171
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Canada | 29 | 35 | 64
  United States | 4 | 2 | 6
  Czechia | 12 | 8 | 20
  Germany | 33 | 31 | 64
  Spain | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Developing AKI, as Defined Per Kidney Disease Improving Global Outcomes (KDIGO) Criteria
Description: Percentage of subjects developing AKI based on Serum Creatinine and/or Urine Output per KDIGO definition
Time Frame: 72 hours
Population: All dosed
Measure: Number; unit: percentage of subjects
Groups:
- RMC-035: RMC-035 is a concentrate (6.0 mg/mL) for solution for infusion for IV administration.
  Dosing was done per kg bodyweight and at Subjects with eGFR ≥60 mL/min/1.73m2 will receive 1.3 mg/kg (per dose) for the first and second dose, followed by 0.65 mg/kg (per dose) for the third, fourth and fifth dose, while subjects with eGFR >30 and <60 mL/min/1.73m2 will receive 0.65 mg/kg (per dose) for all five doses Dosing occurs at time 0 and then after 6, 12, 24 and 48 hours.
  RMC-035: Concentrate for Solution for Infusion
Arm/Group | RMC-035 | Placebo
Number analyzed (Participants) | 89 | 88
percentage of subjects | 50.6 | 39.8

2. Secondary Outcome: Area Under the Curve (AUC) of Serum Creatinine (SCr)
Description: Time-corrected area under the curve (AUC) of serum creatinine calculated as follows:
  The area under the SCr concentration versus time curve following drug administration were calculated using timepoints at Day 1 (12 hour), Day 2 (24 hour), Day 3 (48 hour) and Day 4 (72 hour). The individual log-transformed SCr values were determined, and the AUC (utilizing planned times) were calculated using the right Riemann sum: AUC = 0.5 x SCr(12h) + 0.5 x SCr(24h) + 1 x SCr(48h) + 1 x SCr(72h) The time-corrected AUC (log-scale) was then calculated as AUC/3
Time Frame: 72 hours
Population: all dosed
Measure: Geometric Mean (90% Confidence Interval); unit: log(mg/dL)/day
Arm/Group | RMC-035 | Placebo
Number analyzed (Participants) | 89 | 88
log(mg/dL)/day | 1.13 [1.08 to 1.17] | 0.99 [0.96 to 1.02]

3. Secondary Outcome: Duration of AKI
Description: Duration of AKI defined as the number of days meeting the definition of AKI (KDIGO definition) starting within 72 hours after first dose of IMP until resolution
Time Frame: 90 days
Population: all dosed
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | RMC-035 | Placebo
Number analyzed (Participants) | 89 | 88
Days | 1.5 (2.6) | 1.1 (3.04)

4. Secondary Outcome: Change in SCr Values Over Time
Description: SCr at 12, 24, 48, and 72 hours, respectively, and at Day 7/discharge, Day 30 and Day 90
Time Frame: 90 days
Population: all dosed
Measure: Mean (90% Confidence Interval); unit: mg/dL
Arm/Group | RMC-035 | Placebo
Number analyzed (Participants) | 89 | 88
mg/dL
  12 hours | 0.07 [0.04 to 0.11] | -0.01 [-0.05 to 0.02]
  24 hours | 0.11 [0.06 to 0.15] | 0.01 [-0.04 to 0.05]
  48 hours | 0.08 [0.03 to 0.13] | 0.00 [-0.04 to 0.05]
  72 hours | 0.05 [0.01 to 0.09] | -0.03 [-0.07 to 0.01]
  Day 7 | 0.04 [-0.00 to 0.09] | -0.02 [-0.06 to 0.02]
  Day 30 | -0.00 [-0.04 to 0.04] | 0.01 [-0.02 to 0.05]
  Day 90 | -0.02 [-0.06 to 0.02] | 0.03 [-0.01 to 0.07]

5. Secondary Outcome: Peak Cystatin C Value
Description: Change from baseline of peak cystatin C from baseline to Day 7
Time Frame: 7 days
Population: all dosed
Measure: Mean (90% Confidence Interval); unit: mg/L
Arm/Group | RMC-035 | Placebo
Number analyzed (Participants) | 89 | 88
mg/L | 0.21 [0.16 to 0.26] | 0.11 [0.06 to 0.16]

6. Secondary Outcome: AUC of Cystatin C
Description: Time-corrected AUC of cystatin C for Day 1 to Day 4 (72 hours after first dose of IMP) calculated as follows:
  The area under the cystatin C concentration versus time curve following drug administration were calculated using timepoints at Day 1 (12 hour), Day 2 (24 hour), Day 3 (48 hour) and Day 4 (72 hour). The individual log-transformed cystatin C values were determined, and the AUC (utilizing planned times) were calculated using the right Riemann sum: AUC = 0.5 x cystatin C(12h) + 0.5 x cystatin C(24h) + 1 x cystatin C(48h) + 1 x cystatin C(72h) The time-corrected AUC (log-scale) was then calculated as AUC/3
Time Frame: 72 hours
Population: all dosed
Measure: Geometric Mean (Standard Deviation); unit: log(mg/L)/day
Arm/Group | RMC-035 | Placebo
Number analyzed (Participants) | 89 | 88
log(mg/L)/day | 1.21 (1.28) | 1.09 (1.31)

7. Secondary Outcome: Number of Participants Requiring Renal Replacement Therapy (Dialysis)
Description: Renal replacement therapy (dialysis treatment) required by any participant for any reason
Time Frame: 7 days
Population: all dosed
Measure: Count of Participants; unit: Participants
Arm/Group | RMC-035 | Placebo
Number analyzed (Participants) | 89 | 88
Participants | 1 | 1

8. Secondary Outcome: Number of Days Without Need for Dialysis
Description: Number of days that participants were not requiring dialysis
Time Frame: 90 days
Population: all dosed
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | RMC-035 | Placebo
Number analyzed (Participants) | 89 | 88
Days | 90.0 [90.0 to 90.0] | 90.0 [90.0 to 90.0]

9. Secondary Outcome: Major Adverse Kidney Event (MAKE) - SCr
Description: MAKE at Day 30 and Day 90, defined as death, any dialysis, or ≥25% reduction of eGFR compared to baseline.
  eGFR calculated based on Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation using SCr.
Time Frame: 90 days
Population: all dosed
Measure: Number; unit: percentage of subjects
Arm/Group | RMC-035 | Placebo
Number analyzed (Participants) | 89 | 88
percentage of subjects
  Day 30 | 11.2 | 10.2
  Day 90 | 6.7 | 15.9

10. Secondary Outcome: AKI Within 72 Hours Based on Cystatin C and UO
Description: AKI based on cystatin C and/or urine output (UO)
Time Frame: 72 hours
Population: all dosed
Measure: Number; unit: percentage of subjects
Arm/Group | RMC-035 | Placebo
Number analyzed (Participants) | 89 | 88
percentage of subjects | 48.3 | 40.9

11. Secondary Outcome: AKI Within 7 Days
Description: AKI based on SCr and/or UO criteria, or cystatin C and/or UO criteria
Time Frame: 7 days
Population: all dosed
Measure: Number; unit: percentage of subjects
Arm/Group | RMC-035 | Placebo
Number analyzed (Participants) | 89 | 88
percentage of subjects | 60.7 | 45.5

12. Secondary Outcome: Persistence of AKI
Description: AKI persistence, defined as an AKI (KDIGO definition) developing within 72 hours after first dose of IMP and with a duration of ≥72 hours
Time Frame: 7 days
Population: all dosed
Measure: Number; unit: percentage of subjects
Arm/Group | RMC-035 | Placebo
Number analyzed (Participants) | 89 | 88
percentage of subjects | 18.0 | 14.8

13. Secondary Outcome: Severity of AKI
Description: AKI severity stage 1, 2 or 3 per KDIGO criteria, with 1 being mildest stage and 3 being most severe stage.
  Reference: KDIGO (2012). "Clinical Practice Guideline for Acute Kidney Injury." JOURNAL OF THE INTERNATIONAL SOCIETY OF NEPHROLOGY 2(1).
Time Frame: 7 days
Population: all dosed
Measure: Number; unit: percentage of participants with AKI
Arm/Group | RMC-035 | Placebo
Number analyzed (Participants) | 89 | 88
percentage of participants with AKI
  Stage 1 | 43.8 | 53.8
  Stage 2 | 50.0 | 38.5
  Stage 3 | 6.3 | 7.7

14. Secondary Outcome: Change in Urine Albumin to Creatinine Ratio (UACR) and Urine Protein to Creatinine Ratio (UPCR)
Description: Post-baseline changes in UACR and UPCR at Day 4, Day 30, and Day 90
Time Frame: 90 days
Population: Data were not collected.
Groups:
- RMC-035: RMC-035 is a concentrate (6.0 mg/mL) for solution for infusion for IV administration.
  Dosing will be based on renal function at Day -1: Subjects with eGFR ≥60 mL/min/1.73m2 will receive 1.3 mg/kg (per dose) for the first and second dose, followed by 0.65 mg/kg (per dose) for the third, fourth and fifth dose, while subjects with eGFR >30 and <60 mL/min/1.73m2 will receive 0.65 mg/kg (per dose) for all five doses Dosing occurs at time 0 and then after 6, 12, 24 and 48 hours.
  RMC-035: Concentrate for Solution for Infusion
Arm/Group | RMC-035 | Placebo
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Pharmacokinetics of RMC-035 (AUC)
Description: AUC(0-24) of RMC-035 concentrations in plasma (Day 3)
Time Frame: 4 days
Population: all dosed
Measure: Mean (Standard Deviation); unit: h*ug/mL
Arm/Group | RMC-035
Number analyzed (Participants) | 89
h*ug/mL | 14.63 (12.314)

16. Secondary Outcome: Pharmacokinetics of RMC-035 (Cmax)
Description: Cmax of RMC-035 concentrations in plasma Day 3
Time Frame: 7 days
Population: all dosed
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | RMC-035
Number analyzed (Participants) | 89
ug/mL
  eGFR>=60: number analyzed (Participants) | 55
  eGFR>=60 | 12.59 (25.046)
  eGFR<60: number analyzed (Participants) | 34
  eGFR<60 | 10.62 (3.989)

17. Secondary Outcome: Presence of Anti-drug Antibodies (ADA)
Description: Presence of ADA at Day 1 (pre-surgery), Day 30, and Day 90; positive samples
Time Frame: 90 days
Population: all dosed
Measure: Count of Participants; unit: Participants
Arm/Group | RMC-035 | Placebo
Number analyzed (Participants) | 89 | 88
Participants | 6 | 3

18. Secondary Outcome: Characteristics of ADA (Cross-reactivity)
Description: Characteristics of ADA developed at Day 30 and Day 90 with regards cross-reactivity with endogenous alpha-1-microglobulin (A1M)
Time Frame: 90 days
Population: all dosed
Measure: Count of Participants; unit: Participants
Arm/Group | RMC-035 | Placebo
Number analyzed (Participants) | 89 | 88
Participants | 0 | 0

19. Secondary Outcome: Peak SCr Value
Description: Change from baseline of peak SCr from baseline to Day 7
Time Frame: 7 days
Population: all dosed
Measure: Mean (90% Confidence Interval); unit: mg/dL
Arm/Group | RMC-035 | Placebo
Number analyzed (Participants) | 89 | 88
mg/dL | 0.27 [0.22 to 0.32] | 0.15 [0.10 to 0.20]

20. Secondary Outcome: Major Adverse Kidney Event (MAKE) - Cystatin C
Description: MAKE at Day 30 and Day 90, defined as death, any dialysis, or ≥25% reduction of eGFR compared to baseline.
  eGFR calculated based on Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation using Cystatin C.
Time Frame: 90 days
Population: all dosed
Measure: Number; unit: percentage of subjects
Arm/Group | RMC-035 | Placebo
Number analyzed (Participants) | 89 | 88
percentage of subjects
  Day 30 | 19.1 | 22.7
  Day 90 | 16.9 | 27.3

21. Secondary Outcome: Major Adverse Kidney Event (MAKE) - SCr and Cystatin C
Description: MAKE at Day 30 and Day 90, defined as death, any dialysis, or ≥25% reduction of eGFR compared to baseline.
  eGFR calculated based on Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation using SCr and Cystatin C.
Time Frame: 90 days
Population: all dosed
Measure: Number; unit: percentage of subjects
Arm/Group | RMC-035 | Placebo
Number analyzed (Participants) | 89 | 88
percentage of subjects
  Day 30 | 14.6 | 13.6
  Day 90 | 11.2 | 22.7

22. Secondary Outcome: Change in Serum Cystatin C Values Over Time
Description: Cystatin C measurement in serum at 12, 24, 48, and 72 hours, respectively, and at Day 7/discharge, Day 30 and Day 90
Time Frame: 90 days
Population: all dosed
Measure: Mean (90% Confidence Interval); unit: mg/L
Arm/Group | RMC-035 | Placebo
Number analyzed (Participants) | 89 | 88
mg/L
  12 hours | -0.15 [-0.19 to 0.11] | -0.26 [-0.29 to -0.22]
  24 hours | -0.04 [-0.09 to -0.00] | -0.14 [-0.18 to -0.10]
  48 hours | 0.04 [-0.00 to 0.09] | -0.03 [-0.08 to 0.02]
  72 hours | 0.07 [0.03 to 0.12] | -0.00 [-0.05 to 0.04]
  Day 7 | 0.05 [-0.01 to 0.10] | -0.01 [-0.06 to 0.04]
  Day 30 | 0.10 [0.05 to 0.14] | 0.12 [0.07 to 0.16]
  Day 90 | 0.10 [0.05 to 0.16] | 0.14 [0.08 to 0.19]

ADVERSE EVENTS:
Time Frame: TEAEs (Treatment Emergent Adverse Events): 72 hours after last administration of study intervention, up to 90 days in total.
Description: For non-serious Adverse Events, TEAEs are presented, ie any AE that occurred after the initial IMP administration through 72 hours (inclusive) after the final IMP administration.
  For SAEs, all are presented as per standard definition.
Arm/Group | RMC-035 | Placebo
All-Cause Mortality (participants affected / at risk) | 1/89 | 2/88
Serious Adverse Events (participants affected / at risk) | 20/89 | 15/88
Other Adverse Events (participants affected / at risk) | 75/89 | 64/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RMC-035 (N=89) | Placebo (N=88)
Cerebellar infarction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Embolic cerebral infarction (Nervous system disorders) | 1 | 1
Hemiparesis (Nervous system disorders) | 1 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 1
Status epilepticus (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Arterial haemorrhage (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 5 | 0
Venous haemorrhage (Vascular disorders) | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2
Blood bilirubin increased (Investigations) | 1 | 0
Blood fibrinogen decreased (Investigations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 4 | 0
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1 | 0
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 2 | 2
Cardiac tamponade (Cardiac disorders) | 2 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Low cardiac output syndrome (Cardiac disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RMC-035 (N=89) | Placebo (N=88)
Atrial fibrillation (Cardiac disorders) | 16 | 25
Tachycardia (Cardiac disorders) | 9 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 9 | 13
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 7
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 5
Chills (General disorders) | 27 | 2
Oedema peripheral (General disorders) | 8 | 8
Pyrexia (General disorders) | 11 | 2
Blood creatinine increased (Investigations) | 6 | 1
Haemoglobin decreased (Investigations) | 5 | 0
Anaemia (Blood and lymphatic system disorders) | 17 | 18
Thrombocytopenia (Blood and lymphatic system disorders) | 13 | 8
Leukocytosis (Blood and lymphatic system disorders) | 7 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 | 12
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Procedural pain (Injury, poisoning and procedural complications) | 11 | 9
Nausea (Gastrointestinal disorders) | 19 | 8
Vomiting (Gastrointestinal disorders) | 6 | 3
Hypotension (Vascular disorders) | 10 | 9
Hypertension (Vascular disorders) | 8 | 4
Acute kidney injury (Renal and urinary disorders) | 11 | 11
Delirium (Psychiatric disorders) | 9 | 4
Confusional state (Psychiatric disorders) | 5 | 1

LIMITATIONS AND CAVEATS:
Study was stopped prematurely for futility following Data Monitoring Committee (DMC) recommendation.

The early termination lead to smaller numbers than planned, and that not all outcome measures were analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-10-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT05126303/Prot_002.pdf
  • Statistical Analysis Plan (2023-08-30): https://cdn.clinicaltrials.gov/large-docs/03/NCT05126303/SAP_003.pdf